CLINICAL TRIAL: NCT06583070
Title: Cohort Study of SABR Combined With Targeted Therapy and Anti-PD-1 Versus Targeted Therapy and Anti-PD-1 for Recurrent or Metastatic Renal Cell Carcinoma Patients
Brief Title: SABR Combined With Targeted Therapy and Anti-PD-1 for Recurrent or Metastatic Renal Cancer
Acronym: COSTAR
Status: Recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Collaborators: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: COSTAR-001
Record Dates: First submitted 2024-08-24; First posted 2024-09-03 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-09

CONDITIONS: Radiation Therapy; Metastatic Renal Cancer; Recurrent Renal Cell Cancer
Keywords: SBRT; Metastatic Renal Cancer; Recurrent Renal Cell Cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Radiotherapy; Immunotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RT group: In conjunction with targeted and immunotherapy, administer radiation therapy to achieve as complete coverage as possible of all identifiable primary and metastatic lesions.
  Interventions: Radiation: Radiation therapy; Drug: Targeted and immunotherapy
- Control group: Targeted and immunotherapy
  Interventions: Drug: Targeted and immunotherapy

INTERVENTIONS:
Radiation: Radiation therapy — Administer radiation therapy to achieve as complete coverage as possible of all identifiable primary and metastatic lesions in conjunction with targeted and immunotherapy
  Groups: RT group
Drug: Targeted and immunotherapy — Targeted and immunotherapy

SUMMARY:
Renal cancer ranks seventh in incidence among men and sixth among women in the Beijing area, with Peking University First Hospital treating over 1,000 kidney cancer patients annually. Once recurrence or metastasis occurs, the prognosis is poor, with median progression times of 1-2 years after first-line systemic therapy (targeted therapy combined with immunotherapy). Enhancing local control of lesions is key to improving overall survival. Combining local radiotherapy with systemic treatment may be one approach to address this issue. Currently, Stereotactic Ablative Radiotherapy (SABR) enables precise tumor ablation and can activate the body's immune response. Studies show that the one-year local control rate after SABR exceeds 90%. Preliminary research by the applicant has shown that the combination of drug therapy and SABR for recurrent metastatic renal cancer can extend progression-free survival beyond two years, with earlier intervention leading to more significant survival improvements. This study aims to evaluate the efficacy and safety of combining SABR with targeted and immunotherapy for recurrent metastatic renal cancer through a multicenter, bidirectional cohort design, exploring new therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed renal cancer; diagnosed with recurrent or metastatic renal cancer via PET/CT or other whole-body imaging.
* Evaluated by the radiation oncology and imaging departments as having at least one lesion amenable to radiation therapy.
* Planning to undergo or currently receiving first-line or second-line targeted therapy combined with immunotherapy.
* Voluntarily agrees to participate in the study and signs an informed consent form.
* Male or female, aged ≥18 years (inclusive).
* Expected survival of ≥12 weeks.
* At least one measurable lesion as per the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* European Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate cardiac, bone marrow, liver, and renal function.
* Willing and able to comply with the study procedures and follow-up schedule.

Exclusion Criteria:

* Extensive, multiple metastases;
* Presence of central nervous system metastases and/or carcinomatous meningitis.
* Toxicity from previous treatments not yet recovered to grade 0-1 (excluding grade 2 alopecia);
* Other severe, uncontrollable co-morbid conditions that could affect protocol compliance or confound interpretation of results, including active opportunistic or severe progressive infections, uncontrolled diabetes, uncontrolled hypertension, cardiovascular diseases (defined as New York Heart Association Class III or IV heart failure, second-degree or higher heart block, myocardial infarction within the last 12 months, unstable arrhythmias or angina, stroke within the last 6 months), or pulmonary diseases (interstitial pneumonia, obstructive pulmonary disease, and symptomatic bronchospasm history), deep vein thrombosis or pulmonary embolism within the last 6 months;
* Diagnosed with other malignancies within 5 years prior to enrollment, except:
* Localized low-risk prostate cancer (defined as stage ≤T2b, Gleason score ≤7, and PSA ≤20ng/mL at diagnosis, who have undergone curative treatment with no recurrence of prostate-specific antigen);
* Malignancies treated with a curative intent that are considered cured, including but not limited to adequately treated thyroid cancer, cervical carcinoma in situ, basal or squamous cell skin cancer, or ductal carcinoma in situ of the breast treated with surgery;
* Pregnant or breastfeeding women;
* Positive HIV test result;
* Active hepatitis B or C infection;
* Active tuberculosis;
* Any other conditions, metabolic abnormalities, physical examination or laboratory findings that in the investigator's judgment might indicate an unsuitability for the study drug, could interfere with the interpretation of study results, or place the patient at high risk if they participate in the study;
* Estimated insufficient compliance with the clinical study.

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically confirmed renal cancer; diagnosed with recurrent or metastatic renal cancer via PET/CT or other whole-body imaging.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival 2, PFS2 | 2 year
  Progression Free Survival 2 (PFS2) is defined as the time from the start of treatment to the point where, despite the emergence of new lesions and continuation of the original systemic therapy, local radiotherapy is used to intervene on new lesions. Subsequently, due to the emergence of additional new lesions or progression of existing lesions, a change in systemic therapy becomes necessary. Alternatively, it also includes situations where a new lesion appears and cannot be treated with radiotherapy, necessitating a change in the original systemic therapy plan.

SECONDARY OUTCOMES:
Progression free survival 1, PFS1 | 2 year
  Defined as the time from the start of treatment to the first progression.
Overall survival, OS | 2 year
  Defined as the time from the start of treatment to death.
Objective response rate，ORR | six months.
  Defined as CR (Complete Response) + PR (Partial Response), representing the best response achieved at any time.
Disease control rate，DCR | six months.
  Defined as CR + PR + SD (Stable Disease), maintained for at least six months.
Adverse Reactions | 2 year
  Evaluated using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 to assess treatment-related adverse reactions.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality